CLINICAL TRIAL: NCT02333461
Title: Study to Evaluate Botanicals for Mechanisms Related to Appetite and Fat Metabolism in Healthy, Overweight and Obese Individuals
Brief Title: Evaluation of Botanicals for Mechanisms Related to Appetite and Fat Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Access Business Group (Industry)
Collaborators: Radiant Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BURN CURB POM-1
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — whole grape extract; Prunus armeniaca extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): 333 mg capsule comprised of silicified microcrystalline cellulose, magnesium stearate, modified cellulose gum, silicon dioxide, dextrose, corn starch, and caramel color. Consumed as six capsules once daily (total of 2 g/day) with the morning meal for a period of seven days.
  Interventions: Dietary Supplement: Placebo
- Apple (Experimental): 333 mg capsule comprised of apple peel extract (115:1, standardized to 80% polyphenol and 5% phlorizin). Consumed as six capsules once daily (total of 2 g/day) with the morning meal for a period of seven days.
  Interventions: Dietary Supplement: Apple
- Grape (Experimental): 333 mg capsule comprised of grape extract (8000:1, standardized to 75% total polyphenol, 50% oligomeric proanthocyanidin). Consumed as six capsules once daily (total of 2 g/day) with the morning meal for a period of seven days.
  Interventions: Dietary Supplement: Grape
- Red Raspberry (Experimental): 333 mg capsule comprised of red raspberry leaf extract (4:1, standardized to 6% ellagic acid). Consumed as six capsules once daily (total of 2 g/day) with the morning meal for a period of seven days.
  Interventions: Dietary Supplement: Raspberry
- Apricot/Nectarine (Experimental): 333 mg capsule comprised of apricot/nectarine extract (40:1, standardized to 50% polyphenol).
  Interventions: Dietary Supplement: Apricot/Nectarine

INTERVENTIONS:
Dietary Supplement: Placebo — Participants were randomly assigned to receive one of four botanical interventions or placebo.
  Arms: Placebo
Dietary Supplement: Apple — Participants were randomly assigned to receive one of four botanical interventions or placebo.
  Arms: Apple
Dietary Supplement: Grape — Participants were randomly assigned to receive one of four botanical interventions or placebo.
  Arms: Grape
Dietary Supplement: Raspberry — Participants were randomly assigned to receive one of four botanical interventions or placebo.
  Arms: Red Raspberry
Dietary Supplement: Apricot/Nectarine — Participants were randomly assigned to receive one of four botanical interventions or placebo.
  Arms: Apricot/Nectarine

SUMMARY:
Excess caloric consumption, particularly from inexpensive, energy dense foods that are high in fat and refined carbohydrates, is a major driver of the global obesity epidemic. Dietary supplements that promote reduced intake of energy dense foods and/or impact the absorption and metabolism of fat and carbohydrates in the body can be used to help consumers control their weight. We identified two separate mechanistic approaches to target these effects.

Diacylglycerol acyltransferase-1 (DGAT-1) is an enzyme involved in the formation of dietary fat into circulating triglycerides within the body. Once dietary fat is digested and absorbed, the resulting fatty acids are re-esterified into triglycerides. Inhibition of DGAT-1 results in delayed and decreased re-esterification of dietary fats into circulating triglycerides. It is hypothesized that this effect may lead to decreased deposition of excess dietary fat as adipose tissue, possibly due to increased fatty acid oxidation in the enterocytes.

Ghrelin is a hormone that is known to stimulate appetite in humans. When calorie dense fatty foods are sensed in the stomach, ghrelin is acylated and activated via ghrelin O-acyltransferase (GOAT). The activation step attaches a medium chain fatty acid to the ghrelin molecule that enables it to transmit a signal in the brain that triggers eating and fat storage in adipose tissue. Interfering with the GOAT pathway will inhibit ghrelin activation and possibly diminish food intake and lipid storage. This concept is supported by animal studies in which weight gain in a high fat diet model is prevented when GOAT is inhibited.

Our objective was to determine whether botanicals demonstrating in vitro DGAT-1 and GOAT inhibition have similar mechanistic effects in the human body. Based on the results of this study, prototype formulas may be developed and clinically- tested for outcomes related to weight management.

DETAILED DESCRIPTION:
Excess caloric consumption, particularly from inexpensive, energy dense foods that are high in fat and refined carbohydrates, is a major driver of the global obesity epidemic. Dietary supplements that promote reduced intake of energy dense foods and/or impact the absorption and metabolism of fat and carbohydrates in the body can be used to help consumers control their weight. We identified two separate mechanistic approaches to target these effects.

Diacylglycerol acyltransferase-1 (DGAT-1) is an enzyme involved in the formation of dietary fat into circulating triglycerides within the body. Once dietary fat is digested and absorbed, the resulting fatty acids are re-esterified into triglycerides. Inhibition of DGAT-1 results in delayed and decreased re-esterification of dietary fats into circulating triglycerides. It is hypothesized that this effect may lead to decreased deposition of excess dietary fat as adipose tissue, possibly due to increased fatty acid oxidation in the enterocytes.

Ghrelin is a hormone that is known to stimulate appetite in humans. When calorie dense fatty foods are sensed in the stomach, ghrelin is acylated and activated via ghrelin O-acyltransferase (GOAT). The activation step attaches a medium chain fatty acid to the ghrelin molecule that enables it to transmit a signal in the brain that triggers eating and fat storage in adipose tissue. Interfering with the GOAT pathway will inhibit ghrelin activation and possibly diminish food intake and lipid storage. This concept is supported by animal studies in which weight gain in a high fat diet model is prevented when GOAT is inhibited.

Ghrelin levels are positively associated with stress, sleep deprivation, and caloric restriction. Weight loss induced by exercise does not have the same positive association with ghrelin levels that caloric restriction alone has. Ghrelin levels are influenced by diet composition, however, the results vary considerably between trials.

Over 160 botanical extracts from our internal ingredient library were screened at a single concentration for inhibition of both DGAT-1 and GOAT. Botanicals that were identified as having at least 75% activity were then titrated to identify those with IC50 values < 25 g/ml or less. We narrowed our list of viable ingredients by looking at those with activity in both the DGAT-1 and GOAT in vitro enzyme bioassay models. The top performing botanicals were then evaluated in a cellular model for DGAT-1 inhibition. Those with the highest inhibition activity in this model were considered lead candidates. A preliminary literature search was conducted and the final filter included factors such as cost and regulatory acceptability which results in the four ingredients being tested in the current clinical protocol.Our objective was to determine whether these four ingredients have similar mechanistic effects in the human body.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese (BMI of 25-35 kg/m2) men and women.
* Participant must be 18-70 years of age.
* Considered healthy with no evidence of chronic diseases.
* Willing to maintain a consistent diet and exercise pattern throughout the duration of the study.
* Willing to consume a dairy and egg-based fat challenge meal twice, at start and end of study (V2 & V3).

Exclusion Criteria:

* History of allergic reaction to fruit, dairy or egg products.
* Current smoker or history of tobacco use within the past year.
* Use of dietary supplements within 1 week prior to Visit 2 and unwilling to refrain from use through the duration of the trial. Supplements include any vitamins, minerals, and herbal products, including herbal drinks.
* Use of fish oil supplements within the past 8 weeks.
* Consumption of fatty fish one or more times per week within the past 8 weeks (e.g., mackerel, salmon, trout, canned albacore tuna, sardines, haddock, cod, hake, halibut, shrimp, sole, flounder, perch, black bass, swordfish, oysters, Alaskan king crab).
* Presence of cardiovascular disease, cancer, diabetes mellitus, inflammatory bowel disease, lactose intolerance, or any other chronic health condition identified from the findings of the interview.
* History of gastric bypass or other surgery that physically alters the gastrointestinal tract.
* Blood pressure greater > 140 mm Hg systolic or > 90 mm Hg diastolic during seated, resting measurement on two consecutive occasions during visit 1.
* Fasting serum triglycerides > 200 mg/dl.
* Use of lipid lowering medications or dietary supplements.
* Use of blood pressure lowering medications or dietary supplements.
* Use of Coumadin, aspirin, or other medications that influence hemostasis.
* Daily use of low dose (< 81 mg) aspirin is allowed.
* Use of antibiotics within the past week.
* Chronic or therapeutic use of antacids, H2 agonists, and proton pump inhibitors.
* Use of selective serotonin reuptake inhibitors, monoamine oxidase inhibitors, and/or any other drug with vasoconstricting properties.
* Pregnant or lactating women, or women of child-bearing potential unwilling to use a medically approved form of birth control.
* History, in the past year, of current abuse of drugs or alcohol, or intake > 14 alcoholic beverages per week.
* Participation in another clinical trial within 28 days of enrollment into the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Serum triglyceride response (area under the curve = AUC) following consumption of a standardized high fat meal challenge. | Six hours
Plasma acylated ghrelin response (AUC) following consumption of a standardized high fat meal challenge | Three hours

SECONDARY OUTCOMES:
Maximum concentration (Cmax) for serum triglycerides following consumption of a standardized high fat meal challenge | Six hours
Time to maximum concentration (Tmax) for serum triglycerides following consumption of a standardized high fat meal challenge | Six hours
Cmax for plasma acylated ghrelin following consumption of a standardized high fat meal challenge | Three hours
Tmax for plasma acylated ghrelin following consumption of a standardized high fat meal challenge | Three hours

REFERENCES:
- [Derived] Velliquette RA, Grann K, Missler SR, Patterson J, Hu C, Gellenbeck KW, Scholten JD, Randolph RK. Identification of a botanical inhibitor of intestinal diacylglyceride acyltransferase 1 activity via in vitro screening and a parallel, randomized, blinded, placebo-controlled clinical trial. Nutr Metab (Lond). 2015 Aug 6;12:27. doi: 10.1186/s12986-015-0025-2. eCollection 2015. PMID 26246845